CLINICAL TRIAL: NCT01983514
Title: Intranasal (Optinose Bidirectional Nose-to-brain Device) Versus Intravenous Slow Infusion of Oxytocin - a Randomized, Placebo- Controlled Double-blind, Double-dummy 4-period Cross-over Study in Healthy Adult Volunteers Evaluating Brain Functional Magnetic Resonance Imaging Changes, Cognitive Response, Heart Rate Variability, Plasma Pharmacokinetics and Saliva Concentration After Single-dose Oxytocin 8 or 24 International Units (IU) Intranasally or 1 IU as Slow Intravenous Infusion
Brief Title: Effects of Intranasal Administration of a Single Dose of Oxytocin Using a Novel Device in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OptiNose AS (Industry)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: SMR-2727
Record Dates: First submitted 2013-10-30; First posted 2013-11-14 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Male Adults
Keywords: oxytocin; fMRI; social cognition; heart rate variability; pupillometry; eye tracking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 international unit (IU) intravenous oxytocin (Active Comparator): Using a double-dummy design participants will be administered 1 IU oxytocin (mixed in 200 ml 0.9% sodium chloride) slow infusion with varying infusion rate over 20 minutes and placebo delivered with the OptiNose Breath Powered Bi-Directional liquid device. Subject to pilot data this may be increased to 2 IU oxytocin (mixed in 200 ml 0.9% sodium chloride) and the infusion time/rate may change to best match the pharmacokinetic profile of intranasally administered oxytocin.
  Interventions: Drug: 1 IU intravenous oxytocin
- Placebo (Placebo Comparator): Using a double-dummy design participants will be administered Placebo delivered with the OptiNose Breath Powered Bi-Directional liquid device and placebo delivered intravenously (0.9% sodium chloride 200 ml slow infusion for 20 minutes)
  Interventions: Drug: Placebo
- 8IU intranasal oxytocin (Experimental): Using a double-dummy design participants will be administered 8IU oxytocin liquid delivered with the OptiNose Breath Powered Bi directional liquid device and IV placebo (0.9% sodium chloride, 200 ml slow infusion for 20 minutes)
  Interventions: Drug: 8IU intranasal oxytocin
- 24IU intranasal oxytocin (Experimental): Using a double-dummy design participants will be administered 24IU oxytocin liquid delivered with the OptiNose Breath Powered Bi directional liquid device and IV placebo (0.9% sodium chloride, 200 ml slow infusion for 20 minutes)
  Interventions: Drug: 24 IU intranasal oxytocin

INTERVENTIONS:
Drug: 8IU intranasal oxytocin
  Arms: 8IU intranasal oxytocin
Drug: 24 IU intranasal oxytocin
  Arms: 24IU intranasal oxytocin
Drug: 1 IU intravenous oxytocin
  Arms: 1 international unit (IU) intravenous oxytocin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Oxytocin (OT) is a small, naturally occurring peptide currently in clinical use to stimulate lactation in breastfeeding women. The intranasal administration of OT has recently attracted attention as a potential novel treatment in several psychiatric disorders including autism. However, given the anatomy of the nasal cavity, the current design of nasal sprays would be expected to provide an inadequate delivery of medication to the areas of the nasal cavity where direct transport into the brain via the olfactory nerve could potentially occur. OptiNose has developed an intranasal delivery device that provides improved reproducibility of nasal delivery, improved deposition to the upper posterior regions of the nasal cavity where the olfactory nerve innervates the nasal cavity.

The primary objective of this study is to identify any differences between single dose 8 or 24 international units (IU) oxytocin delivered intranasally with the optimised OptiNose device and 1 IU oxytocin administered as slow intravenous infusion in healthy volunteers. This will be measured in terms of brain activity as measured with functional magnetic resonance imaging (fMRI), performance on cognitive tests, and physiological markers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male subjects aged 18 to 35 years inclusive.
* Subjects must be in good general health, as determined by the investigator.
* Subject's pre-study physical examination, vital signs and electrocardiogram (ECG) are normal or do not show any clinically significant abnormalities as determined by the investigator. Vital signs must not have any clinically significant deviations outside of the following ranges when measured sitting after 5 minutes rest:

  1. Heart rate: 40 to 90 beats per minute
  2. Systolic blood pressure (BP): 90 to 140 mmHg
  3. Diastolic BP: 50 to 90 mmHg
  4. Oral temperature: 36.0 to 37.5°C
  5. Respiratory rate: 12 - 18 breaths per minute
* Body Mass Index (BMI) of 18.5 - 29.9 kg/m2 (both inclusive)
* Subjects must be able to communicate well with the Investigator, to understand and comply with the requirements of the study, and understand and sign the written informed consent
* Provision of written informed consent.

Exclusion Criteria:

An ear, nose and throat (ENT) specialist will inspect the noses of all individuals who enter the study.

In order to participate in the study subjects must not meet any of the following exclusion criteria;

* Individuals showing major septal deviation or a significantly altered nasal epithelium.
* Participants with evidence of previous nasal disease, surgery, and dependence on inhaled drugs.
* Individuals with current significant nasal congestion due to common colds.
* Subjects with a clinically relevant history of significant hepatic, renal, endocrine, cardiac, nervous, psychiatric, gastrointestinal, pulmonary, haematological or metabolic disorder.
* Subjects with current or history of, any clinically significant disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Subject is taking any regular prescribed or over-the-counter (OTC) medications including vitamin supplements and herbal remedies. There must be at least 14 days between stopping these products and the first dose of study medication).
* Systemic illness requiring treatment within 2 weeks prior to Study Day 1.
* History of significant drug or alcohol abuse (as per a self-report measure / instrument; World Health Organisation criteria/Alcohol use disorders identification test/Drug use disorders identification test). Subjects with a positive screen for alcohol or drugs of abuse at screening/admission will be excluded from participation in the study.
* Self-reported significant psychiatric conditions.
* Any abnormal laboratory values outside normal range, and which is clinically significant as deemed by investigator.
* Full scale intelligence quotient (IQ) < 75 (due to the prerequisite ability to complete self report measures).
* Known allergic reactions or hypersensitivity to any component of the study medication in the nasal spray, such as E216, E218 and chlorobutanol hemihydrate.
* Participation in any (other) clinical trial with an investigational medicinal product or medical device within 3 months prior to randomisation.
* Current evidence of any mental or physical disorder or collaboration attitude which, in the judgment of the investigator makes the subject unsuitable for enrolment, and/or may interfere with the study evaluations or affect subject's safety.
* Subjects with any metal implants.
* Subjects with claustrophobia.
* Other unspecified reasons that, in the opinion of the Investigator or the sponsor make the subject unsuitable for enrolment.
* Subjects with female partners of child-bearing potential must use an adequate form of contraception prior to entry into the study until three months following the post-study medical visit. Subjects must not have a partner who is either pregnant or breastfeeding for the duration of the study. Adequate contraception is defined as the usage by the female partner of any form of hormonal contraception or intra-uterine device (which should be established prior to the start of the study) plus usage by one of the partners of an additional spermicide- containing barrier method of contraception.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Aim 1a: Brain activity | 30 minutes after oxytocin/placebo administration
  Scanning procedures for functional magnetic resonance imaging (fMRI) will include a functional scan during a social cognition task and structural connectivity during rest
Aim 1b: Performance on a social cognition test | 45 mins after oxytocin/placebo administration
  Participants will complete a task evaluating emotional expressions (either happy expressions, fear expressions or neutral expressions). These stimuli are identical to those published previously by Leknes et al., (2012).
Aim 1c: Heart rate variability | 20 minutes after oxytocin placebo administration
  Electrocardiogram data will be collected to assess heart rate variability, a measure of cardiac autonomic function.
Aim 1d: Eyetracking | 20 minutes after oxytocin placebo administration
  An eyetracking device will measure eyegaze and pupillometry.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of oxytocin | 5 minutes prior to oxytocin/placebo administration
  Blood will be collected to assess levels of oxytocin present in peripheral blood to measure PK profile of 8 and 24 international units (IU) oxytocin delivered with OptiNose device and of 1 IU oxytocin after slow intravenous (IV) infusion.
Plasma concentration of cortisol | 20 minutes before fMRI procedure
  Blood will be drawn at various intervals for the pharmacokinetic analysis of plasma cortisol.
Oxytocin levels in saliva | 20 prior to fMRI procedure
  Saliva will be collected for pharmacokinetic analysis of oxytocin and cortisol in saliva.
Cortisol levels in saliva | 20 minutes prior to fMRI procedure
  Saliva will be collected for pharmacokinetic analysis of oxytocin and cortisol in saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Ole A Andreassen, MD, Principal Investigator — University of Oslo
Locations (1):
- Norwegian Centre for Mental Disorders Research (NORMENT), KG Jebsen Centre for Psychosis Research - TOP Study, Oslo, Norway

REFERENCES:
- [Background] Leknes S, Wessberg J, Ellingsen DM, Chelnokova O, Olausson H, Laeng B. Oxytocin enhances pupil dilation and sensitivity to 'hidden' emotional expressions. Soc Cogn Affect Neurosci. 2013 Oct;8(7):741-9. doi: 10.1093/scan/nss062. Epub 2012 May 29. PMID 22648957
- [Derived] Quintana DS, Westlye LT, Alnaes D, Rustan OG, Kaufmann T, Smerud KT, Mahmoud RA, Djupesland PG, Andreassen OA. Low dose intranasal oxytocin delivered with Breath Powered device dampens amygdala response to emotional stimuli: A peripheral effect-controlled within-subjects randomized dose-response fMRI trial. Psychoneuroendocrinology. 2016 Jul;69:180-8. doi: 10.1016/j.psyneuen.2016.04.010. Epub 2016 Apr 22. PMID 27107209
- [Derived] Quintana DS, Westlye LT, Rustan OG, Tesli N, Poppy CL, Smevik H, Tesli M, Roine M, Mahmoud RA, Smerud KT, Djupesland PG, Andreassen OA. Low-dose oxytocin delivered intranasally with Breath Powered device affects social-cognitive behavior: a randomized four-way crossover trial with nasal cavity dimension assessment. Transl Psychiatry. 2015 Jul 14;5(7):e602. doi: 10.1038/tp.2015.93. PMID 26171983
- See also: Click here for more information about NORMENT: Norwegian Centre for Mental Disorders Research — http://www.med.uio.no/norment/english/